CLINICAL TRIAL: NCT04888039
Title: Therapeutic and Support Oncologic Medical Care Evaluation in Patients With Multiple Myeloma in West-Occitanie Region. Factors Influencing Medical Care and Predictive and Prognostic Impact.
Brief Title: Follow-up of Patients With Multiple Myeloma in the West-Occitanie Region "Living With a Myeloma in West-Occitanie"
Acronym: VAMOS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Takeda (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0482; N° ID RCB: 2020-A03527-32 (Registry Identifier: Numéro ID RCB)
Record Dates: First submitted 2021-05-04; First posted 2021-05-17 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Real life; Health care pathways; Quality of life
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: quality of life questionnaires (EORTC QLQ-C30 ; EORTC QLQMY20 ; EQ-5D-5L ; Cohen's stress scale) — Excepted the delivery of quality of life questionnaires (a maximum of 5 times during the course of treatment) specific to this study, only the data available during the course of patient care will be collected.
  The quality of life questionnaires and the perceived stress questionnaire will be given to patients :
  * At diagnosis (before starting 1st line of treatment),
  * after the induction phase (before autologous transplantation for patients who will be transplanted),
  * after the consolidation phase,
  * after the maintenance phase : 1 year and 2 years after the start of the maintenance.

SUMMARY:
Actually very few real life data are available for patients with multiple myeloma (MM), whereas they're playing a more and more important role in health care decisions. Treatments choice for medical care of patient with MM depends of their age, their general status, their eligibility to high dose treatment (autograft), and also based on cytogenetic risk (standard/high risk). Therapeutic strategies are multiple and based on drugs associations including proteasome inhibitors, immuno-modulators and monoclonal antibodies.

Therapeutic medical care objective is to improve quality and response duration through more effective induction schemas, systematic consolidation for patients who have undergone high dose therapy and/or maintenance treatment, ensuring patients safety and well-being in the health care pathway.

Quality of life evaluation has to take in consideration disease outcome and secondary effects impact from treatments prescribed for MM.

With clinical trials, new therapeutic strategies are proposed with innovative drugs but participants are selected and do not represent all patients with MM. Therefore, there is a large gap between clinical trials and real life data.

That's why the CHU Toulouse intends to set up a prospective cohort to evaluate the health care pathway of patients with MM in West-Occitanie region and studies impact of treatments prescribed on the disease and on the patients' quality of life.

With this research, standard of care practices for patients with MM will be followed, prognostic scores and clinical trials results will be validated in real life, impact of outpatient support procedure will be assessed (AMA procedure) and sociodemographic/quality of life data will be available for research teams.

DETAILED DESCRIPTION:
Primary objective :

Describe health care pathways of patients with MM living in West Occitanie according to socio-demographic patients' caracteristics, their comorbidities and their initial disease severity. These pathways will be described until the patients' death if the death occurs before the end of their follow-up in this study.

Secondary objectives :

* The best response at each line of therapy
* The progression free survival and overall survival
* Quality of life of patients with MM along their health care pathway
* Second primary malignancy and neuropathy grade 3 or more occurrence during patients'care
* Socio-demographic, clinic and biology factors identification to predict response to treatments, progression free survival, overall survival and quality of life.

Study size calculation :

With the hypothesis of 80% of patients informed about the study will agree to participate and will accept to have their health care data collected, and with 500 to 550 patients' medical files presented each year for MM care to West Occitanie multidisciplinary committee meeting (approximately 400 different patients), a 5-years recruitment period will lead to 1600 patients enrollment.

This size will be able to generate enough precisions for descriptive analyses. Indeed, as example, with a percentage of 50%, conservative situation to estimate percentages, expected precision should be more or less 2.5% according to Clopper-Pearson exact method.

Precision of more or less 5% should be also obtained for sub-groups of 400 persons.

ELIGIBILITY:
Inclusion Criteria:

* Patient living in the West-Occitanie region
* Patient with a diagnosis of symptomatic multiple myeloma (Rajkumar et al, Lancet Oncology 2014)

Exclusion Criteria:

* Patient opposed to this research
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a diagnosis of symptomatic multiple myeloma and living in the west-Occitanie region.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2031-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Treatment lines and procedures followed by the patients | 5 to 10 years
  Different treatment lines and procedures followed by the patients with drugs involved, number of cycles performed in each treatment phase (induction, consolidation, maintenance) and for each therapeutic line
Transplants | 5 to 10 years
  Transplants carrying out
Treatments discontinuation | 5 to 10 years
  Reasons for treatments administered discontinuation
Therapeutic medical care description | 5 to 10 years
  Supportive care and the type of care set up
Unconventional alternative medicine | 5 to 10 years
  Use and description of unconventional alternative medicine
Outpatient support structure | 5 to 10 years
  Support from an outpatient support structure (AMA)

SECONDARY OUTCOMES:
Best response (BR) | 5 to 10 years
  BR evaluated according to IMWG criteria at each treatment line. This takes into account the MRD as part of the response criteria since this date.
Progression-free Survival (PFS) | 5 to 10 years
  Time between date of first intake of treatment until 1st progression according to the IMWG criteria or until death if it occurs before progression
PFS after the second therapeutic line | 5 to 10 years
  Time between date of 1st dose of treatment until 2nd progression according to the IMWG criteria or until death if it occurs before the 2nd progression.
Overall Survival (OS); | 5 to 10 years
  Time between date of first intake of treatment and death from any cause.
Quality of life (QOL) during the treatment course | 5 to 10 years
  QOL assessed by the EORTC questionnaires QLQ-C30, QLQMY20 and EQ-5D-5L, at the start of treatment then at the end of induction and consolidation periods and once a year for patients undergoing maintenance for the first 2 lines of treatment.
Second primary cancers (SPC) and grade 3 and higher neuropathies | 5 to 10 years
  -SPC and grade 3 and higher neuropathies (depending on the applicable version of the CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Aurore PERROT, MD, Principal Investigator — IUCT-Oncopole - Toulouse University Hospital
Locations (1):
- IUCT-Oncopole - Toulouse University Hospital, Toulouse, West-Occitanie, France

IPD SHARING:
Plan to Share IPD: Undecided